CLINICAL TRIAL: NCT04922047
Title: Safety and Efficacy Study of Tislelizumab Alone and in Combination With Bacille Calmette-Guérin (BCG) in High-Risk Non-Muscle-Invasive Bladder Cancer (NMIBC) Patients, a Prospective Open Single-site Trial（TACBIN-01）
Brief Title: Safety and Efficacy Study of Tislelizumab in Combination With BCG in HR-NMIBC Patients (TACBIN-01)
Acronym: TACBIN-01
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: BeiGene (Industry); Huidu Shanghai Medical Sciences Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2021-041; BGB-A317-2002-IIT (Other: Beigene)
Record Dates: First submitted 2021-06-06; First posted 2021-06-10 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Urinary Bladder Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Antineoplastic Agents; Urinary Bladder Diseases; Tislelizumab Antineoplastic Agents, Immunological
Keywords: bladder carcinoma; BCG; PD-1
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Urinary Bladder Diseases | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Intravenous tislelizumab / Intravesical BCG (Experimental): Drug: tislelizumab / BCG
  Tislelizumab 200 mg administered by intravenous infusion every 3 weeks in first year and continue to second year based on physician choose. BCG 120 mg induction therapy administered via intravesical instillation (once weekly for 6 weeks). BCG induction therapy is followed by maintenance therapy (once weekly for 3 weeks at months 3, 6, 12, 18, 24m).
  Other Name: BGB-A317
  Interventions: Drug: tislelizumab and BCG

INTERVENTIONS:
Drug: tislelizumab and BCG — Tislelizumab 200 mg administered by intravenous infusion every 3 weeks in first year and continue to second year based on physician choose. BCG 120 mg induction therapy administered via intravesical instillation (once weekly for 6 weeks). BCG induction therapy is followed by maintenance therapy (once weekly for 3 weeks at months 3, 6, 12, 18, 24m).

SUMMARY:
This study is a single-arm, open-label, single-center study to assess the safety of tislelizumab with BCG, and to obtain the preliminary efficacy results in subjects who have been diagnosed with high-risk NMIBC without prior BCG treatment.

DETAILED DESCRIPTION:
An estimated 130,000 new cases were diagnosed with bladder cancer in China each year. About 75-85% of them are NMIBC. The standard care for high risk (HR) NMIBC is intravesicular BCG instillation. Despite BCG treatment, 40% of patients will eventually experience a recurrence, which is associated with a poorer prognosis.

This is a single center Phase I safety and efficacy study of tislelizumab with BCG treatment. The study will determine the safety of administering tislelizumab at 200mg iv q3w in conjunction with intravesicular BCG treatment in HR NMIBC patients who was treatment-naïve or BCG naïve, but underwent TURBT to remove all resectable disease (residual CIS acceptable) within 6 weeks and confirm absence of muscle invasion.

BCG installation was the stander treatment for HR NMIBC. Despite BCG treatment, 40% of patients will eventually experience a recurrence, which is associated with a poorer prognosis. It was reported that BCG increased antigen expression and cytokine release from tumor cells, leading to immune cell (e.g. CD4+ and CD8+T cells, NK, macrophages) recruitment and immune-mediated cytotoxicity (indirect effect). PD-L1 expression intravesicular is found to be extremely abundant in the tumor tissue in patients failing BCG treatment. Which may inhibit the T cell to eliminate cancer cells. Based on these data, a combination of tislelizumab with BCG may be effective in preventing recurrence of NMIBC.

The 6 subjects will be treated at a dose of 200 mg tislelizumab with 120 mg BCG to explode safety for the combination though observing DLT within 28days. If no safety issues are present, we will carry out multi-cohort Phase II study（TACBIN-02）

ELIGIBILITY:
Inclusion Criteria:

* Adult man and women, 18-75 years old ECOG PS 0-1
* Life expectancy ≥1year
* Any high risk non muscle invasive urothelial carcinoma histologically confirmed defined on the TURBT within 6weeks as any of the following :
* T1 tumor and/or
* High grade (WHO 2004) and/or Grade 3 (WHO1973) and/or
* Carcinoma in situ (CIS)
* Underwent TURBT to remove all resectable disease (residual CIS acceptable) within 6 weeks before recruitment and confirm absence of muscle invasion. The restagingTURBT is acceptable, but the interval between the two TURBTs is 2-6 weeks;
* Absence of metastasis in pelvis, abdomen, or chest, as confirmed by a negative baseline computed tomography (CT) or magnetic resonance imaging (MRI) scan no more than 3m prior to the first study treatment
* BCG-naïve defined as：
* Chemotherapy failure but BCG naïve: patients who have received at least six of eight induction doses of chemotherapy（including immediate single instillation）have a high risk of recurrence within 1 year; but have not received BCG perfusion in the bladder;
* Treatment-naïve: patients who have not received prior intravesical chemotherapy or BCG, but who previously received but stopped chemotherapy or BCG more than 3 years before study entry are eligible
* Adequate hematologic and organ function, as defined by the following laboratory results obtained within 14 days prior to the first dose:
* white blood cell (WBC) counts ≥ 3.0× 109/L
* absolute neutrophil count (ANC) ≥1.5 ×109/L
* Platelet count ≥ 75 ×109/L
* Hemoglobin ≥ 9.0 g/dL
* Serum albumin ≥ 30g/L
* aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase(ALP) ≤2.5 × the upper limit of normal (ULN)
* Serum bilirubin ≤1.0 × ULN
* Partial thromboplastin time (PTT)/Prothrombin Time (PT) ≤1.5 × ULN or international normalized ratio (INR) <1.7 × ULN
* Calculated creatinine clearance ≥ 30 mL/min (Cockcroft-Gault formula)
* Female participants of childbearing potential have a negative urine or serum pregnancy test before recruitment. Female or male must be willing to use an adequate method of contraception during the treatment period and for at least 5 months after the last dose of tislelizumab
* Patient is willing and able to sign a written informed consent document and comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits, and examinations including follow-up.

Exclusion Criteria:

* Muscle-invasive, locally advanced non-resectable, or lymph node positive, or metastatic urothelial carcinoma; previous or accompanied by upper urinary tract urothelial carcinoma (UTUC)
* There are pathological variants or non-urothelial cancer components in the very high risk of NMIBC
* T1 high-grade (HG/G3) combined with urothelial carcinoma of the prostate urethra
* Pathological tissue specimens with lymphovascular infiltration or special type of urothelial carcinoma after TURBT*

  *Special types of urothelial carcinoma: adenoid differentiation, squamous differentiation, neuroendocrine differentiation, plasma cell-like changes and micropapillary changes, etc.
* Prior treatment with CD137 agonists or immune checkpoint-blockade therapies, including anti-CD40, anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* The diagnosis of HR NMIBC was followed by induction intravesical chemotherapy, but immediate single instillation (within 24 hours after surgery) was allowed before the pathological results were not clear. The drugs include mitomycin, pirarubicin, doxorubicin, epirubicin, CHPT or gemcitabine;
* Treatment with anti-cancer therapy including systemic immunostimulatory agents (including but not limited to INF, IL-2any), chemotherapy, radiation therapy, or hormonal therapy or any other investigational agent.
* Any unresolved toxicity (CTCAE grade 2 or above) from previous anti-cancer therapy.
* Active autoimmune disease that has required systemic treatment in the past 2 years, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease and so on.
* Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days before first dose. The use of inhaled or low-dose (e.g., ≤10 mg/day prednisone) corticosteroids is allowed.
* Known HIV, active Hepatitis B or C infection or tuberculosis.
* Infections ≥ 3 grade within 4 weeks, including but not limited to severe urinary tract infection, severe pneumonia, infectious complications, bacteremia intravenous antibiotic therapy or hospitalization patients receiving therapeutic oral or IV antibiotics within 1 weeks prior to the first dose are not eligible.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Allergy or hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the tislelizumab or BCG formulation
* Prior allogeneic stem cell or solid organ transplant
* Major surgical procedure other than for diagnosis within 4 weeks prior to the first dose or anticipation of need for a major surgical procedure during the study
* Patients who have any of the following cardiac conditions:
* Poorly controlled diabetes (after treatment with glycosylated hemoglobin [HbA1c]> 8%);
* Poorly controlled High blood pressure evaluated by the investigator (blood pressure >160mmHg/100mmHg);
* Cardiac insufficiency (including left ventricular ejection fraction [LVEF] <50%), myocardial infarction within the past 6 months, arrhythmia or unstable angina that cannot be well controlled by medication.
* Pulmonary embolism, chronic obstructive pulmonary disease, interstitial lung disease or clinically significant lung function test abnormalities; oother conditions that the treating physicians believe may endanger the health of the patients by their participation in this clinical trial.
* Administration of a live, attenuated vaccine within 4 weeks prior to first dose, during treatment or within 8 weeks following the last dose of tislelizumab Note: Seasonal vaccines for influenza are generally inactivated vaccines and are allowed.
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, in situ cervical cancer, prostate cancer without evidence of PSA progression or carcinoma in situ such as the following: gastric, prostate, cervix, colon, melanoma, or breast for example.
* Have a mental illness, restricted or incapable of civil conduct, and a known history of psychotropic drug abuse. It may increase the risk of participating in the research, or interfere with the results of the research, and patients who the researcher believes are not suitable for participating in this research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days of single infusion
  Safety

SECONDARY OUTCOMES:
Event Free Survival (EFS) rate at 24 months | approximately 24 months
  efficacy
Progression free survival (PFS) rate at 36 months | approximately 36 months
  efficacy
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | approximately 24 months
  Safety

OTHER OUTCOMES:
Biomarker (Tissue, liquid biopsy) | approximately 24 months
  Explorative outcome

CONTACTS AND LOCATIONS:
Overall Officials: Wei XUE, MD, PHD, Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Investigator Link — https://zhangruiyun4337.haodf.com/